CLINICAL TRIAL: NCT01371214
Title: Maintaining Independence in Alzheimer's Disease
Brief Title: Preventing Loss of Independence Through Exercise (PLIÉ) - Pilot
Acronym: PLIÉ-pilot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Deborah Barnes, Associate Professor, Psychiatry and Epidemiology & Biostatistics, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 10-04080-023906
Record Dates: First submitted 2011-06-07; First posted 2011-06-10 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Dementia
Keywords: exercise; exercise movement techniques; activities of daily living
MeSH Terms: conditions — Dementia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): PLIÉ exercise program 30-45 minutes, 2-3 days/week for 18 weeks followed by 18 weeks of usual care (20-minutes of chair-based exercises 2-5 days/week).
  Interventions: Behavioral: PLIÉ (Preventing Loss of Independence through Exercise)
- Group 2 (Active Comparator): Usual care (20 minutes of chair-based exercises 2-5 days/week) for 18 weeks followed by the PLIÉ exercise program 30-45 minutes/day, 2-3 days/week for 18 weeks.
  Interventions: Behavioral: PLIÉ (Preventing Loss of Independence through Exercise)

INTERVENTIONS:
Behavioral: PLIÉ (Preventing Loss of Independence through Exercise) — Integrative exercise program that incorporates elements of Eastern and Western exercise traditions to target the muscles and movements needed to help individuals with mild to moderate dementia maintain functional status and independence.

SUMMARY:
The primary goal of this study is to perform a 36-week pilot study with a cross-over design to study the safety and efficacy of a novel integrative exercise program called PLIÉ (Preventing Loss of Independence through Exercise). PLIÉ integrates elements of Eastern and Western exercise traditions and is specifically designed to target the muscles and movements needed to help individuals with mild-to-moderate dementia maintain physical function and independence.

ELIGIBILITY:
Inclusion Criteria - Primary Participant:

* Current participant in the Irene Swindells Center for Adult Day Services in San Francisco, CA
* Recommended by Swindells staff
* mild-to-moderate dementia
* caregiver consent

Inclusion Criteria - Caregiver:

* Provide care to primary participant in the Irene Swindells Center for Adult Day Services in San Francisco, CA
* can provide information about the primary participant's physical functioning, behaviors, falls, quality of life and own level of stress.

Exclusion Criteria - Primary Participant:

* major current psychiatric illness (e.g., schizophrenia, bipolar disorder)
* life expectancy < 1 year (e.g., metastatic cancer)
* inability to assent to study procedures

Exclusion Criteria - Caregiver:

* Any major neurologic disease (e.g., dementia, stroke, Parkinson's disease, ALS)
* major current psychiatric illness (e.g., schizophrenia, bipolar disorder)
* life expectancy < 1 year (e.g., metastatic cancer)
* evidence of cognitive impairment
* inability to consent to study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in physical function (participant) | Baseline, 18 weeks, 36 weeks
  Participant's physical function will be assessed with the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) scale (Galasko 1997). The ADCS-ADL is a 78-point scale that assesses functional ability in 23 daily activities based on informant report. It is the standard measure for assessment of functional status in AD treatment trials.
Change in quality of life (participant) | Baseline, 18 weeks, 36 weeks
  Quality of life will be assessed with the Quality of Life Scale in Alzheimer's Disease (QOL-AD), which is a brief, 13-item measure that obtains input from both the individual and the caregiver (Logsdon 1999). Scores may range from 13-52 points.
Change in functional health and well-being (participant) | Baseline, 18 weeks, 36 weeks
  Functional health and well-being will be assessed with the SF-36v2, which assesses function in eight domains and provides physical and mental component summary scores that may range from 0 to 70 (Stewart 1989). The SF-36v2 is typically administered directly to participants. However, we also will ask caregivers to answer questions on behalf of participants and will compare their answers to assess congruence. Data collected will help to determine if this measure is suitable for a larger trial.
Change in number of falls (participant) | Baseline, 18 weeks, 36 weeks
  Participant's falls will be assessed based on caregiver report.
Change in fall-related self-efficacy (participant) | Baseline, 18 weeks, 36 weeks
  Fall-related self-efficacy will be assessed with the Falls Efficacy Scale (FES), which is a 10-item scale that has been validated in individuals with cognitive impairment (Hauer 2010).
Change in physical performance (participant) | Baseline, 18 weeks, 36 weeks
  Physical performance will be assessed with the Short Physical Performance Battery (SPPB), which was developed by the National Institute on Aging to provide an objective tool for evaluating lower extremity functioning in older adults. The test includes repeated chair stands, tandem balance testing and 8' walking speed (Guralnik 1994).
Change in cognitive function (participant) | Baseline, 18 weeks, 36 weeks
  Cognitive function will be assessed with the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog) (Rosen 1984), which is the most commonly used primary outcome measure in AD treatment trials. It is an 80-point scale that includes direct assessment of learning (word list), naming (objects), following commands, constructional Praxis (figure copying), ideational Praxis (mailing a letter), orientation (person, time, place), recognition memory and remembering test instructions.
Compliance (participant) | Baseline, 18 weeks, 36 weeks
  Participant compliance will be determined based on % of exercise classes attended from baseline to 18 weeks and from 18-36 weeks.
Adverse events (participant) | Baseline, 18 weeks, 36 weeks
  Number of adverse events from baseline to 18 weeks and from 18 weeks to 36 weeks will be monitored through biweekly telephone calls with caregivers.
Change in dementia-related behaviors (participant) | Baseline, 18 weeks, 36 weeks
  Participant's dementia-related behaviors will be assessed with the Neuropsychiatric Inventory (NPI), which is a 144-point informant-based questionnaire that assesses 12 behavioral domains common in dementia including frequency, severity and impact on caregiver distress (Cummings 1997).

SECONDARY OUTCOMES:
Change in functional health and well-being (caregiver) | Baseline, 18 weeks, 36 weeks
  Caregivers will be asked about the functional health and well-being of themselves as well as participants using the SF-36v2, which assesses function in eight domains and provides physical and mental component summary scores that may range from 0 to 70 (Stewart 1989).
Change in burden (caregiver) | Baseline, 18 weeks, 36 weeks
  Caregiver burden will be assessed with the Caregiver Burden Inventory (CBI), which is a 96-point scale that includes 24 items and 5 domains (Novak 1989).

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Barnes, PhD, MPH, Principal Investigator — University of California, San Francisco; Margaret Chesney, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Irene Swindells Center for Adult Day Services, Institute on Aging, San Francisco, California, United States

REFERENCES:
- [Result] Barnes DE, Mehling W, Wu E, Beristianos M, Yaffe K, Skultety K, Chesney MA. Preventing loss of independence through exercise (PLIE): a pilot clinical trial in older adults with dementia. PLoS One. 2015 Feb 11;10(2):e0113367. doi: 10.1371/journal.pone.0113367. eCollection 2015. PMID 25671576
- [Result] Wu E, Barnes DE, Ackerman SL, Lee J, Chesney M, Mehling WE. Preventing Loss of Independence through Exercise (PLIE): qualitative analysis of a clinical trial in older adults with dementia. Aging Ment Health. 2015;19(4):353-62. doi: 10.1080/13607863.2014.935290. Epub 2014 Jul 14. PMID 25022459